CLINICAL TRIAL: NCT02854306
Title: Psycho-sensorial Mindfulness and Top-down Control : Mindfulness Program for Obese Patients in Preparation to Bariatric Surgery
Brief Title: Mindfulness in Preparation to Bariatric Surgery
Acronym: PConscience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 38RC12.215
Record Dates: First submitted 2016-07-13; First posted 2016-08-03 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Obesity
Keywords: Bariatric surgery; Mindfulness; Obese
MeSH Terms: conditions — Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgery (Active Comparator): Obese patient without mindfulness program in parallel.
  Interventions: Procedure: Bariatric surgery
- Surgery with mindfulness program (Active Comparator): Obese patient following a mindfulness program in parallel.
  Interventions: Procedure: Bariatric surgery

INTERVENTIONS:
Procedure: Bariatric surgery — With mindfulness programm
Procedure: Bariatric surgery — Without mindfulness programm

SUMMARY:
Mindfulness is a common practice already widely used, that has shown benefits in terms of psychological and physical health. It is about learning or learn again to be self present and aware to the environment, across breathing, sensations, emotions and thought centering exercises, in the present moment without any judgement.

The goal is to evaluate the efficacy of "mindfulness" versus an active control group in bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients: over 18 years
* Patients suffering from morbid obesity (BMI ≥ 40 kg/m²), or severe obesity (BMI ≥ 35 kg/m²) associate with at least a comorbidity likely to be improved by surgery
* Patient revised in second-line after the failure of a well conducted medical treatment, nutritional, dietetic and psychotherapeutic during 6 to 12 months : absence of enough weight loss or absence of maintain of weight loss
* Absence of any psychiatric counter-argument

Exclusion Criteria:

* Subjects responding to inclusion criteria of the French National Authority for Health
* Subjects without agoraphobia, or obsessive-compulsive disorder, in post-traumatic stress disorder, alcohol or drugs dependant, without psychotic disorders, major depressive disorder, or suffering from anti-social personality disorder
* Patient registered for social security
* Free, signed and informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2014-11-14 (Actual)

PRIMARY OUTCOMES:
Psychometric evaluation | About 15 minutes
  Tool : SBC-20 - Scale of Body Connexion
Psychometric evaluation | About 15 minutes
  Tool : TAS-20 - The twenty-item Toronto Alexithymia Scale
Psychometric evaluation | 15 minutes
  Tool : BAQ-18- Body Awareness Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Yves Benhamou, Professor, Principal Investigator — Grenoble Hospital University
Locations (1):
- UniversityHospitalGrenoble, La Tronche, France

REFERENCES:
- [Background] Breslin KT, Reed MR, Malone SB. An holistic approach to substance abuse treatment. J Psychoactive Drugs. 2003 Apr-Jun;35(2):247-51. doi: 10.1080/02791072.2003.10400006. PMID 12924747
- [Background] Cserjesi R, Luminet O, Poncelet AS, Lenard L. Altered executive function in obesity. Exploration of the role of affective states on cognitive abilities. Appetite. 2009 Apr;52(2):535-9. doi: 10.1016/j.appet.2009.01.003. PMID 19260167
- [Background] Heatherton TF, Baumeister RF. Binge eating as escape from self-awareness. Psychol Bull. 1991 Jul;110(1):86-108. doi: 10.1037/0033-2909.110.1.86. PMID 1891520
- [Background] Jon-Kabat-Zinn. (2009) Au cœur de la tourmente, la pleine conscience : MBSR, la réduction du stress basée sur la mindfulness, Bruxelles, De Boeck, coll. Carrefour des Psychothérapies
- [Background] Grossman P, Niemann L, Schmidt S, Walach H. Mindfulness-based stress reduction and health benefits. A meta-analysis. J Psychosom Res. 2004 Jul;57(1):35-43. doi: 10.1016/S0022-3999(03)00573-7. PMID 15256293
- [Background] Keng SL, Smoski MJ, Robins CJ. Effects of mindfulness on psychological health: a review of empirical studies. Clin Psychol Rev. 2011 Aug;31(6):1041-56. doi: 10.1016/j.cpr.2011.04.006. Epub 2011 May 13. PMID 21802619
- [Background] Karason K, Molgaard H, Wikstrand J, Sjostrom L. Heart rate variability in obesity and the effect of weight loss. Am J Cardiol. 1999 Apr 15;83(8):1242-7. doi: 10.1016/s0002-9149(99)00066-1. PMID 10215292
- [Background] Leahey T.M., Crowther J. H., Irwin S.R. (2008) A cognitive-behavioral mindfulness group therapy intervention for the treatment of binge eating in bariatric surgery patients. Cognitive and Behavioral Practice, 15(4), p.364-375.
- [Background] Lutz A, McFarlin DR, Perlman DM, Salomons TV, Davidson RJ. Altered anterior insula activation during anticipation and experience of painful stimuli in expert meditators. Neuroimage. 2013 Jan 1;64:538-46. doi: 10.1016/j.neuroimage.2012.09.030. Epub 2012 Sep 19. PMID 23000783
- [Background] Lutz A, Slagter HA, Dunne JD, Davidson RJ. Attention regulation and monitoring in meditation. Trends Cogn Sci. 2008 Apr;12(4):163-9. doi: 10.1016/j.tics.2008.01.005. Epub 2008 Mar 10. PMID 18329323
- [Background] Mobbs O, Crepin C, Thiery C, Golay A, Van der Linden M. Obesity and the four facets of impulsivity. Patient Educ Couns. 2010 Jun;79(3):372-7. doi: 10.1016/j.pec.2010.03.003. Epub 2010 Apr 18. PMID 20399590
- [Background] Moeller FG, Barratt ES, Dougherty DM, Schmitz JM, Swann AC. Psychiatric aspects of impulsivity. Am J Psychiatry. 2001 Nov;158(11):1783-93. doi: 10.1176/appi.ajp.158.11.1783. PMID 11691682
- [Background] Nederkoorn C, Smulders FT, Havermans RC, Roefs A, Jansen A. Impulsivity in obese women. Appetite. 2006 Sep;47(2):253-6. doi: 10.1016/j.appet.2006.05.008. Epub 2006 Jun 19. PMID 16782231
- [Background] Praissman S. Mindfulness-based stress reduction: a literature review and clinician's guide. J Am Acad Nurse Pract. 2008 Apr;20(4):212-6. doi: 10.1111/j.1745-7599.2008.00306.x. PMID 18387018
- [Background] Price CJ, Wells EA, Donovan DM, Rue T. Mindful awareness in body-oriented therapy as an adjunct to women's substance use disorder treatment: a pilot feasibility study. J Subst Abuse Treat. 2012 Jul;43(1):94-107. doi: 10.1016/j.jsat.2011.09.016. Epub 2011 Nov 25. PMID 22119181
- [Background] Taylor GJ. Alexithymia: concept, measurement, and implications for treatment. Am J Psychiatry. 1984 Jun;141(6):725-32. doi: 10.1176/ajp.141.6.725. PMID 6375397
- [Background] Van Strien T, Engels RC, Van Leeuwe J, Snoek HM. The Stice model of overeating: tests in clinical and non-clinical samples. Appetite. 2005 Dec;45(3):205-13. doi: 10.1016/j.appet.2005.08.004. Epub 2005 Oct 20. PMID 16242809
- [Background] Waller G, Babbs M, Wright F, Potterton C, Meyer C, Leung N. Somatoform dissociation in eating-disordered patients. Behav Res Ther. 2003 May;41(5):619-27. doi: 10.1016/s0005-7967(03)00019-6. PMID 12711268
- [Background] Weineland S, Arvidsson D, Kakoulidis TP, Dahl J. Acceptance and commitment therapy for bariatric surgery patients, a pilot RCT. Obes Res Clin Pract. 2012 Jan-Mar;6(1):e1-e90. doi: 10.1016/j.orcp.2011.04.004. PMID 24331170
- [Background] Wiser S, Telch CF. Dialectical behavior therapy for Binge-Eating Disorder. J Clin Psychol. 1999 Jun;55(6):755-68. doi: 10.1002/(sici)1097-4679(199906)55:63.0.co;2-r. PMID 10445865